CLINICAL TRIAL: NCT06912334
Title: Investigation of the Effects of Transcutaneous Vagus Nerve Stimulation on Fibromyalgia. A Double Blind, Sham-controlled Randomized Clinical Trial
Brief Title: Transcutaneous Vagus Nerve Stimulation on Fibromyalgia- Double-blind, Sham-controlled Randomized Clinical Trial
Acronym: TVNS- Fibro
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Martina Rekatsina, Assisitant Professor Of Anaesthesiology, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 566/21-020-2024
Record Dates: First submitted 2025-03-06; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Transcutaneous Vagus Nerve Stimulation on Fibromyalgia
Keywords: vagus nerve; vagus nerve stimulation; tVNS; transcutaneous vagus nerve stimulation; fibromyalgia; FM; double blind; sham controlled; randomized clinical trial; pain; depression; sleep disorders; fatigue; fibro fog; 2016 revised FM ACR Classification Criteria
MeSH Terms: conditions — Fibromyalgia; Pain; Depression; Sleep Wake Disorders; Fatigue

STUDY DESIGN:
Intervention Model Description: A double blind, sham-controlled randomized clinical trial
  * 1st group: Standard pharmacological Treatment according to EULAR + active tVNS, 30min/session, 7 days/week for 2 weeks (14 sessions total)
  * 2nd group: Standard pharmacological Treatment according to EULAR + sham tVNS, 30min/session, 7 days/week for 2 weeks (14 sessions total)
  * Regarding the standard pharmacological treatment we will follow a stepwise approach according to the EULAR (European League Against Rheumatism) recommendations.
Who Masked: Participant, Investigator
Masking Description: Randomization and Blinding Subjects that meet the inclusion criteria will be randomized to either the active (group 1) or the sham tVNS group (group 2). The assignment will be predetermined by a randomized assignment list, created prior to the enrollment of the first subject by an investigator from the Pain Clinic team who is not directly involved in subject treatment. The list will be created with randomization.org. There will be concealed allocation of treatment assignment such that investigators involved in subject screening, consent, and clinical scoring will be blinded to treatment condition.
  The subjects will be informed that they have a 50-50 chance of receiving either active or sham stimulation. Additionally, the assigned clinical evaluators will remain blinded to the stimulation condition. A medical provider not involved in the study will make the allocation of each patient according to the number.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active tVNS group (Active Comparator): 1st group Standard pharmacological Treatment according to EULAR + active tVNS, 30min/session, 7 days/week for 2 weeks (14 sessions total) Regarding the standard pharmacological treatment we will follow a stepwise approach according to the EULAR (European League Against Rheumatism) recommendations. The patients will be randomized by using randomization.org
  Interventions: Device: tVNS
- sham tVNS group (Sham Comparator): 2nd group Standard pharmacological Treatment according to EULAR + sham tVNS, 30min/session, 7 days/week for 2 weeks (14 sessions total) Regarding the standard pharmacological treatment we will follow a stepwise approach according to the EULAR (European League Against Rheumatism) recommendations. The patients will be randomized by using randomization.org
  Interventions: Device: tVNS

INTERVENTIONS:
Device: tVNS — tVNS L is a battery-driven electrical stimulator connected to an ear electrode which is positioned over the skin of the cymba conchae. Thus, auricular vagal stimulation will be applied using the typical ear electrodes of the tVNS® L device. tVNS will be applied over the left branch for safety reasons. For sham auricular tVNS, the anodal electrode will be placed over the center of the left ear lobe. The cathode will be placed over the antitragus. This method and these stimulation parameters have been previously used for reliable blinding in other clinical studies. Series of electrical pulses with 250 μs pulse width, 25 Hz frequency, and 28 s inter-burst interval (32 sec on/28 sec off duty cycle) will be applied in each intervention session. Auricular tVNS will be applied at 1mA - 5mA intensity for 30 min per session (1 session per day, 7 consecutive days a week, 14 sessions in total)
  Other Names: NEMOS L tVNS device from the Neuraxon company

SUMMARY:
Stimulation of the vagus nerve, a parasympathetic nerve that controls the digestive, the vascular and immune systems, produces pain relief in various clinical conditions. Transmission via vagal afferents to the nucleus of the solitary tract has been proposed as the primary physiological mechanism that reduces pain intensity following vagal stimulation. Medication is one of the pillars of dealing with chronic pain, with several benefits, but also side effects. Fibromyalgia is an idiopathic chronic pain syndrome with few, effective and safe treatments. However, current research in the field of vagal innervation suggests psychophysiological and electrical ways by which the syndrome may be treated.The chronic pain symptoms of fibromyalgia patients may benefit from vagus nerve stimulation, by normalizing the autonomic and immune system dysfunction that causes their respective symptoms. However, the effects of multiple sessions of transcutaneous vagus nerve stimulation (tVNS) in fibromyalgia have not been evaluated in randomized clinical trials. The hypothesis of our study is to evaluate if the addition of transcutaneous stimulation of the auricular branch of the vagus nerves in patients with fibromyalgia, can lead to better pain control and quality of life. We will offer a 2-week treatment (14 sessions of 30 minutes) in a randomized double-blind controlled trial. The sample of the study, which will be conducted in the pain clinic of the Aretaieion University General Hospital, will be consisted of 120 patients, who will be divided into 2 groups (1st group: standard pharmacological treatment + active tVNS, 2nd group: standard pharmacological treatment + sham tVNS). The study is designed to determine, if standard pharmacological treatment combined with 14 sessions of tVNS is able to improve pain symptomatology in fibromyalgia and all symptoms of this syndrome, by using appropriate scales. This study examines a new and potentially impactful way to address a major public health issue where prevalence is high in given groups, its impact is multidimensional and treatment options are limited. The holistic treatment of chronic pain, including its neurobiological, cognitive, behavioral and psychological components, may become a valuable aid in the completion of the research project, with the ultimate aim of the study being the establishment of non-invasive stimulation of the vagus nerve for the treatment of chronic pain in clinical practice in the future.

DETAILED DESCRIPTION:
Fibromyalgia is a multidimensional disease, as many factors contribute to its development (biological, genetic, psychosocial). As a result, it demands a multifaceted approach, from patient education to pharmacological treatment etc. Regarding the pharmacotherapy, that should be aimed at a mechanism-oriented fashion. [7] Consistent with this approach, centrally acting medications can be effective in fibromyalgia, particularly antidepressants and anticonvulsants, which increase the presence of pain-inhibitory neurotransmitters by facilitating descending pathways and decreasing dorsal horn sensitization, or decreasing systemic hyperexcitability. Clinical trials have failed to conclusively provide overall benefits of specific therapies to treat fibromyalgia. Therefore, current pharmacological treatments for patients suffering from this syndrome are mainly directed to palliate some symptoms, with relevant clinical benefits experienced only by a minority of individuals.

In those treated with pharmacotherapy, a 50% reduction in pain intensity is generally achieved only by 10% to 25%. However, some treatments seem to significantly improve the quality of life of certain FM patients. Only a few drugs have been approved for use in the treatment of FM by the US Food and Drug Administration (FDA), whereas no drug has been approved for this indication by the European Medicines Agency. Thus patients with FM frequently need to be treated on an off-label basis. Currently, only 25% to 40% pain reduction is granted by drugs and meaningful relief occurs in only 40% to 60%, in part due to dose-limiting adverse effects and incomplete drug efficacy. These limitations in clinical practice have led some to hypothesize that a combination of different analgesic drugs acting through different mechanisms may provide superior outcomes compared to monotherapy. Moreover, drugs should be started at low doses and cautiously titrated because severalpatients, either do not tolerate or benefit from drug therapy. Because sleep disturbance, pain and psychological distress are the most amenable to drug therapy, drugs should be chosen to manage the individual's predominant symptoms. Currently, several drugs are frequently used alone or in combination to manage FM symptoms. However, the US FDA indicated for FM only three: two selective serotonin and norepinephrine reuptake inhibitors (SNRIs), duloxetine and milnacipran as well as an anticonvulsant, pregabalin. Although clinical evidence demonstrating the efficacy or effectiveness of opioids analgesics is scanty, these molecules are widely used for the treatment of FM. However, the long-term use of opioids in FM has been discouraged by several medical guidelines. As a result, there comes a need of a new treatment of fibromyalgia syndrome, which will be effective, safe, easily applied, with almost no side effects and low cost. Non-invasive neuromodulation techniques are gaining more and more the interest of the scientific society as regards a variety of medical conditions, such as chronic pain, epilepsy, rheumatoid arthritis. Transcutaneous Vagus Nerve Stimulation (tVNS) is one of these new techniques.

The parasympathetic vagus nerve (10th cranial nerve) innervates multiple internal organs and integrates sensory, motor, and autonomic information by four vagal nuclei. The primary central relay of vagal afferents is the nucleus of the solitary tract in the brainstem, and several branches of this nucleus, project to different brain areas. The myelinated A- and B-fibers of the vagal nerve send somatosensory, motor, and autonomic signals, and the complex system of vagal projections is involved in inflammatory, immune, nociceptive, and emotional processes. A relevant role of the vagal nerve in pain processing is the transmission of peripheral inflammation signals to the central nervous system. Neuromodulatory activity has been identified in areas related to the sensory and emotional processing of pain, such as the insular cortex and the Anterior Cingulate Cortex (ACC), after vagal stimulation, which reveals that the central system of pain processing receives vagal afferences. In 1988 the first human implant of a vagal stimulating device was performed. In 1997, the US Food and Drug Administration (FDA) approved the use of Vagal Nerve Stimulation (VNS) as anadjunctive treatment for medically refractory epilepsy. Vagus nerve stimulation is a FDA-approved treatment for different pathologies. The regulation of the autonomic and immune systems and a specific effect on chemical mediators of inflammation are relevant physiological mechanisms of the VNS.

At the present research study, we will use the 2016 revision to 2010/2011 ACR fibromyalgia diagnostic criteria. The treatment of fibromyalgia is based on a biopsychosocial approach and includes pharmacological and non-pharmacοlogical approaches, according to the EULAR recommendations. However, patients are still reporting high pain scores and increased interference with quality of life.

Considering that the vagus nerve controls pain signals towards the central nervous system and growing evidence of autonomic dysfunction in fibromyalgia in terms of sympathetic hyperactivity, it can be argued that rebalancing the sympathetic- parasympathetic activity via vagal stimulation might reduce the intensity of pain and stabilize the autonomic symptoms of this disease. In addition, an immune system alteration seems to mediate the interaction between the autonomic nervous system and the chronic inflammatory state in fibromyalgia, apparently by the influence of inflammatory cytokines and chemokines. Stimulation of the auricular and cervical branches of the vagus nerve might reduce such inflammatory overactivity via efferent modulation of the activity of the inflammatory processes and hereby reduce pain symptoms. The potential of non-invasive stimulation of the auricular and cervical branches of the vagus nerve in repeated sessions to improve fibromyalgia symptoms has not been evaluated in randomized, sham-controlled clinical studies. Transcutaneous stimulation of the auricular and cervical branches of the vagus nerve (tVNS), are both non-invasive, low-intensity electric stimulation procedures. According to literature, the effectiveness of these non-invasive methods might not differ significantly from the invasive vagus nerve stimulation, while non-invasiveness provides an advantageous safety profile. Since fibromyalgia involves a dysregulation of the autonomic and immune systems, non-invasive tVNS is expected to improve the symptoms of fibromyalgia, including chronic, musculoskeletal, and generalized pain, through modulation of the vegetative and immune systems. The purpose of the proposed double blind placebo controlled randomized clinical trial is to investigate the effect of tVNS in Chronic Pain compared to medication and the future establishment of the given technique in the clinic. The research interest of the scientific community is growing more and more in recent years. However, research in thisfield is still in its infancy stages. At the same time the holistic treatment of chronic pain, including its neurobiological, psychosocial, cognitive and behavioral components, may become a valuable aid-giver in the best completion of the research project. Research question and Aim The hypothesis of our study is to evaluate, if the addition of transcutaneous stimulation of the auricular branch of the vagus nerves in patients suffering with fibromyalgia can lead to better pain control and quality of life. To investigate this, we will offer a 2 week treatment (14 sessions) in a double-sham controlled study.

This study is designed to determine whether the standard pharmacological treatment paired with 14 sessions of tVNS can improve pain symptomatology in fibromyalgia and the whole range of FM symptoms, such as depression, anxiety, fatigue etc. by using appropriate scales as Numerical Rating Scale (NRS), Fibromyalgia Impact Questionnaire (FIQ), Brief Pain Inventory (BPI), Depression and Anxiety Stress Scale (DASS), Materials and Methods (binding+sham) Participants Our population will be comprised of fibromyalgia patients that are originally diagnosed or referred to Aretaieion Pain Clinic. For the diagnosis (or confirmation of diagnosis) we will be using the ACR (American College of Rheumatology) 2016 revised criteria.

The present single center double blind sham-controlled randomized clinical trial will be conducted at the Pain Clinic of Aretaieion University Hospital, National and Kapodistrian University of Athens. Recruitment Methods Investigators may contact (or be contacted by) a potential subject by telephone or email or direct contact to discuss participation in this research protocol. The investigator will provide the subject with all the information contained in the written consent form and at the same time she will answer any questions regarding the research and give the subject sample, time to consider participation in the study, which may require a follow-up phone conversation or an in-person appointment at the Pain Clinic for a brief study enrollment screening visit.

ELIGIBILITY:
Inclusion Criteria

* Women between 18-79 years old
* Women diagnosed with Fibromyalgia according to the ACR 2016 Revised Classification Criteria
* Moderate to high pain intensity according to analog pain scales (above 4 points over 10), for more than 6 months
* Cognitive function sufficient to understand the experiments and follow instructions
* Ability to read and understand all information on the device display.
* Ability to adjust the strength of the stimulation or give feedback regarding their response to the device (feeling tingling/pulsating/pain).
* Ability to comply with the recommended therapy regiment of 30 min per day.
* The ear electrode needs to fit the patient.
* Patients with physical or mental disabilities
* The patient must be able to use the device by themselves or
* The patients' caretaker can operate the device on the patient. In this case the patient --must still be able to give feedback regarding their response to the device

Exclusion Criteria

* Cardiac arrhythmias
* Pregnancy
* Serious mental disorder (dipolar disorder, schizophrenia etc.)
* Prior injury to the vagus nerve
* Individuals with scar tissue that may interfere with the stimulation
* Presence of an electrically or magnetically activated implant

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity and Fibromyalgia symptoms | 2 weeks
  numerical rating scale pain score (NRS) and Brief Pain Inventory (BPI) and Fibromyalgia Symptoms according to 2016 FM ACR Classification Criteria

SECONDARY OUTCOMES:
Fatique | 2 weeks
  NRS scale
Depression | 2 weeks
  DASS
Sleep Disorders | 2 weeks
  Symptom Severity Scale
Fibro Fog | 2 weeks
  Symptom Severity Scale
Fibromyalgia Symptoms | 2 weeks
  FiRST - Fibromyalgia Rapid Screening Tool

CONTACTS AND LOCATIONS:
Locations (1):
- Aretaieion University Hospital, Athens, Greece, Greece